CLINICAL TRIAL: NCT04570839
Title: A Phase 1/2 Study Evaluating the Safety, Tolerability and Preliminary Antitumor Activity of COM701 in Combination With BMS-986207 (Anti-TIGIT Antibody) and Nivolumab in Subjects With Advanced Solid Tumors.
Brief Title: COM701 in Combination With BMS-986207 and Nivolumab in Subjects With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Compugen Ltd (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPG-03-101.
Record Dates: First submitted 2020-09-18; First posted 2020-09-30 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Endometrial Neoplasms; Ovarian Cancer; Solid Tumor; Head and Neck Cancer
Keywords: TIGIT; PVRIG; checkpoint inhibitor; Immune checkpoint; Immuno-oncology; CD226; CD112; CD155; Solid tumor; Ovarian cancer; Endometrial cancer; PVRL2; Basket study; Opdivo; DNAM
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms; Head and Neck Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Sequential dose escalation, followed by an expansion cohort upon determination of the recommended dose for expansion (RDFE) of COM701 in combination with BMS-986207 and nivolumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation Cohorts. (Experimental): Up to 5 sequential dose escalation cohorts of COM701 in combination with fixed doses of BMS-986207 and nivolumab. All study drugs will be administered IV every 4 weeks until a maximum tolerated dose or recommended dose for expansion is identified.
  Interventions: Drug: COM701 in combination with BMS-986207 and nivolumab.
- Cohort 1 Expansion Cohort A (ovarian cancer) (Experimental): Single arm: subjects with platinum resistant/refractory epithelial ovarian cancer, primary peritoneal or fallopian tube cancer will be randomized to receive study treatment with COM701 in combination with BMS-986207 and nivolumab. The study drugs will be administered IV every 4 weeks.
  Interventions: Drug: COM701 in combination with BMS-986207 and nivolumab.
- Cohort 2 Expansion Cohort (endometrial cancer). (Experimental): Single arm: subjects with MSS-endometrial cancer will receive study treatment with COM701 in combination with BMS-986207 and nivolumab. All study drugs will be administered IV every 4 weeks.
  Interventions: Drug: COM701 in combination with BMS-986207 and nivolumab.
- Cohort 3 Expansion Cohort (basket cohort - high PVRL2 tumors). (Experimental): Single arm: subjects with tumor types with high expression of PVRL2 will receive study treatment with COM701 in combination with BMS-986207 and nivolumab. All study drugs will be administered IV every 4 weeks.
  Interventions: Drug: COM701 in combination with BMS-986207 and nivolumab.
- Cohort 4 Expansion Cohort (Head and Neck cancer). (Experimental): Two arms: subjects with head and neck cancer. Equal number of subjects in each of the 2 arms. One arm will enroll subjects who have not previously received treatment with an immune checkpoint inhibitor, the other arm will enroll subjects who have received prior treatment with an immune checkpoint inhibitor.
  All subjects will receive study treatment with COM701 in combination with BMS-986207 and nivolumab. All study drugs will be administered IV every 4 weeks.
  Interventions: Drug: COM701 in combination with BMS-986207 and nivolumab.

INTERVENTIONS:
Drug: COM701 in combination with BMS-986207 and nivolumab. — Study treatment with the 3 drug combination (COM701 in combination with BMS-986207 and nivolumab).

SUMMARY:
This is a phase 1/2 open label sequential dose escalation and cohort expansion study evaluating the safety, tolerability and preliminary antitumor activity of COM701 in combination with BMS-986207 and nivolumab in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This phase 1/2 study evaluates the safety/tolerability, pharmacokinetics and preliminary antitumor activity of COM701 an inhibitor of poliovirus receptor related immunoglobulin domain containing (PVRIG) in combination with BMS-986207 (an inhibitor of TIGIT) and nivolumab in subjects with advanced solid tumors. The study will consist of 2 parts (part 1 - dose escalation and part 2 - dose expansion).

Part 1: escalating doses of COM701 will be combined with fixed doses of BMS-986207 and nivolumab. Upon completion of dose escalation a recommended dose of COM701 in combination with BMS-986207 and nivolumab (3-drug combination) will be determined.

Part 2: subjects will be administered the recommended dose of COM701 in combination with BMS-986207 and nivolumab. Subjects will be enrolled into one of three cohorts based on their cancer type.

Cohort 1: subjects with platinum resistant/refractory ovarian cancer, primary peritoneal or fallopian tube cancer will receive study treatment with the 3-drug combination.

Cohort 2: subjects with MSS- endometrial cancer will receive study treatment with the 3-drug combination.

Cohort 3 (Basket cohort): subjects with tumors that have high expression of a biomarker (PVRL2) will receive study treatment with the 3-drug combination. Subjects with tumor types in cohorts 1, 2 and 4 will not be enrolled into this cohort.

Cohort 4: subjects with HNSCC. This cohort will enroll subjects who have received treatment with an immune checkpoint inhibitor or subjects who have received treatment with chemotherapy but not an immune checkpoint inhibitor. All subjects enrolled in this cohort will receive study treatment with the 3-drug combination.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed, locally advanced or metastatic solid malignancy and has exhausted all available standard therapy or is not a candidate for the available standard therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* During dose escalation - Subjects who received prior therapy with anti-PD-1, anti-PD-L1, anti- CTLA-4, OX-40, CD137, etc., are eligible.

During cohort expansion: All subjects must have measurable disease as defined by RECIST v1.1.

Expansion Cohorts:

* Cohort 1 (subjects with advanced epithelial ovarian, fallopian tube, or primary peritoneal carcinoma)
* Subject must have platinum refractory/resistant ovarian cancer defined as refractoriness to platinum-containing regimen or disease recurrence < 6 months after completion of a platinum-containing regimen
* Cohort 2 (endometrial cancer cohort)
* Subjects with locally advanced or metastatic microsatellite stable endometrial cancer with disease recurrence or progression during or after prior therapy that included platinum-based chemotherapy.
* Subjects must have documented MSS status by an approved test e.g. genomic testing, IHC for mismatch repair proficient.
* Subjects must have received no more than 2 prior systemic cytotoxic therapies; there are no limits to the number of prior endocrine or antiangiogenic regimens
* Cohort 3 (basket cohort, excludes tumor types in cohorts 1 and 2)
* Tumor types with high expression of PVRL2 (determined by central testing).
* Cohort 4 (Head and Neck cancer)
* Histologically confirmed recurrent or metastatic HNSCC (oral cavity, oropharynx, larynx, hypopharynx, nasopharynx, paranasal sinus, nasopharyngeal)
* Cohort 4a - IO naïve. Eligible subjects can be systemic therapy naïve (frontline) or platinum failure.
* Cohort 4b - IO failure. No limitations on the number of prior lines of systemic therapy.

Key Exclusion Criteria:

* Active autoimmune disease requiring systemic therapy in the last 2 years prior to the first dose of COM701.
* Symptomatic interstitial lung disease or inflammatory pneumonitis.
* History of immune-related events that lead to immunotherapy treatment discontinuation.
* Untreated or symptomatic central nervous system (CNS) metastases.

Key Exclusion Criteria For Dose Expansion Cohorts:

* Cohort 1: Prior therapy with an anti-PD-1/PD-L1/2, COM701 (or any inhibitor of PVRIG), anti-TIGIT antibody, anti-CTLA-4 antibody, anti-OX-40 antibody, anti-CD137 antibody.
* Cohort 2: Prior therapy with COM701 (or any inhibitor of PVRIG) or anti-TIGIT antibody. Subjects with MSI-H endometrial cancer are ineligible.
* Cohort 3: Prior therapy with COM701 (or any inhibitor of PVRIG) or anti-TIGIT antibody are ineligible.
* Cohort 4: Subjects who have received prior therapy with COM701 (or any inhibitor of PVRIG), anti-TIGIT antibody, anti-CTLA-4 antibody, anti-OX-40 antibody, anti-CD137 antibody. Subjects in cohort 4a must be IO-naïve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with adverse events on the study. | 2 years.
  The proportion of subjects with any adverse event (AE) per CTCAE v5.0.
The proportion of subjects with adverse events in the 1st cycle during dose escalation within the DLT window (28 days). | Within the DLT window (1st 28 days) of the 1st cycle during dose escalation.
  The proportion of subjects with adverse events meeting the criteria of dose-limiting toxicities (DLTs) in the 1st 28 days of the 1st cycle of study treatment during dose escalation.
The recommended dose for expansion (RDFE) of the combination. | 2 years.
  The dose of COM701 in combination with BMS-986207 and nivolumab for the expansion cohort.
The Area under the curve of COM701 in subjects receiving the 3-drug combination. | 2 years.
  The PK profile of COM701 in combination with BMS-986207 and nivolumab.

SECONDARY OUTCOMES:
The objective response rate of subjects enrolled in cohorts 1-4. | 3 years.
  Objective response rate per RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Lead COM701 ClinInfo, Study Director — Compugen Ltd
Locations (9):
- United States (9):
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins University Oncology Center., Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - START Midwest., Grand Rapids, Michigan
  - Columbia University, New York, New York
  - University of Pittsburgh Cancer Center., Pittsburgh, Pennsylvania
  - The University of Tennessee WEST Cancer Center., Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - The START Center for Cancer Care., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No